CLINICAL TRIAL: NCT02456389
Title: A Randomized Controlled Trial of Perioperative Risk Stratification and Risk-based, Protocol-driven Management in Patients Undergoing Elective Major Cancer Surgery
Brief Title: Perioperative Risk Study
Acronym: PRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-073
Record Dates: First submitted 2015-05-01; First posted 2015-05-28 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Tumors; Primary Neoplasm; Secondary Neoplasm; Surgery
Keywords: Probable cancer; Proven cancer; Elective cancer surgery; Postoperative death; Postoperative complications; Healthcare utilization; Quality of life; Adjuvant therapy; Disease-free survival; Overall survival
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard perioperative management (Active Comparator): Standard postoperative care
  Interventions: Other: Standard postoperative care
- Risk-based, perioperative management (Experimental): Preoperative risk stratification Postoperative risk stratification Risk-based, escalating levels of care Risk-based, escalating levels of monitoring Risk-based, escalating levels of co-management
  Interventions: Other: Preoperative risk stratification; Other: Postoperative risk stratification; Other: Risk-based, escalating levels of care; Other: Risk-based, escalating levels of monitoring; Other: Risk-based, escalating levels of co-management

INTERVENTIONS:
Other: Preoperative risk stratification — Preoperative risk-prediction tool based on patient demographics/co-morbidity and planned procedure
  Arms: Risk-based, perioperative management
Other: Postoperative risk stratification — Postoperative risk-prediction tool based on intraoperative variables
  Arms: Risk-based, perioperative management
Other: Risk-based, escalating levels of care — Postoperative observation in regular unit vs. telemetry unit vs. stepdown unit vs. ICU
  Arms: Risk-based, perioperative management
Other: Risk-based, escalating levels of monitoring — Varying frequencies of vital signs monitoring Varying use of telemetry, pulse oximetry, and early warning system
  Arms: Risk-based, perioperative management
Other: Risk-based, escalating levels of co-management — Varying use of Hospitalist co-management
  Arms: Risk-based, perioperative management
Other: Standard postoperative care — Routine postoperative care, as medically indicated
  Arms: Standard perioperative management

SUMMARY:
The primary objective of this trial is to determine if perioperative risk stratification and risk-based, protocol-driven management leads to a reduction in the rate of death or serious complications compared to standard perioperative management in patients undergoing elective major cancer surgery.

DETAILED DESCRIPTION:
Major cancer surgery is associated with significant rates of postoperative mortality and major morbidity. Postoperative morbidity adversely impacts healthcare utilization, healthcare costs, rates of discharge to home, quality of life, rates of receipt of postoperative anti-neoplastic therapy, disease-free survival, and overall survival. The investigators hypothesize that perioperative risk stratification and risk-based, protocol-driven management (compared to standard perioperative management) will lead to a reduction in 30-day post-operative mortality or major morbidity in patients undergoing major cancer surgery. This is based on our theory that preoperative/postoperative use of newly developed, perioperative risk-prediction tools will help identify patients at increased risk of postoperative death or serious complications that might benefit from risk-based, protocol-driven perioperative management, including escalating levels of care, escalating levels of monitoring, and escalating levels of hospitalist co-management. The set of assessments and interventions in the proposed study are conceptually similar to other "bundled" interventions which have recently been recently tested and demonstrated to reduce perioperative mortality and morbidity.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age > or = 18 years at diagnosis.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2, or 3.
3. Probable (i.e., clinically suspicious) or histologically/cytologically confirmed, primary or recurrent, malignant neoplasm, malignant neuroendocrine tumor, or carcinoma in situ (any stage).
4. Scheduled for curative or palliative major cancer surgery, including:

   * Glossectomy
   * Pharyngectomy
   * Laryngectomy
   * Neck dissection
   * Esophagectomy
   * Lung resection
   * Gastrectomy
   * Pancreatectomy
   * Hepatectomy
   * Colectomy
   * Proctectomy
   * Hysterectomy/Myomectomy
   * Gynecologic reconstruction
   * Prostatectomy
   * Nephrectomy
   * Cystectomy
   * Breast reconstruction
   * Flap reconstruction
5. Scheduled for elective major cancer surgery at Fox Chase Cancer Center within 30 days after First Registration.
6. Ability to understand and willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent document
7. Geographical accessibility and willingness to return to Fox Chase Cancer Center for all preoperative and postoperative study assessments.

EXCLUSION CRITERIA:

1. Clinical or tissue diagnosis of benign neuroendocrine tumor, benign neoplasm, neoplasm of uncertain behavior, or neoplasm of unspecified nature.
2. Use of systemic chemotherapy and/or radiation therapy < 14 days prior to First Registration. Palliative radiation therapy is permitted for irradiating small areas of painful bony metastases that cannot be managed adequately using systemic or local analgesics
3. Any condition that might interfere with the subject's participation in the study, compliance with study requirements, or in the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1456 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of death or serious complications (as defined by American College of Surgeons National Surgical Quality Improvement Program [ACS NSQIP]) | 30-day postoperative period

SECONDARY OUTCOMES:
Rate of death | 30-day postoperative period
Rate of serious complication (as defined by ACS NSQIP) | 30-day postoperative period
Rate of serious/grade 3-4 adverse event (as defined by CTCAE) | 30-day postoperative period
Rate of Clavien-Dindo grade IIIa-V complication (as defined by ACS NSQIP) | 30-day postoperative period
Rate of Clavien-Dindo grade IIIa-V adverse event (as defined by CTCAE) | 30-day postoperative period
Rate of cardiac complications | 30-day postoperative period
Rate of pulmonary complications | 30-day postoperative period
Rate of renal complications | 30-day postoperative period
Rate of wound complications | 30-day postoperative period
Rate of infectious complications | 30-day postoperative period
Rate of return to the operating room | 30-day postoperative period
Rate of primary intensive care unit admission | From date of index surgery to date of hospital discharge, up to 3 months
Rate of secondary intensive care unit admission | From date of index surgery to date of hospital discharge, up to 3 months
Length of stay | From date of index surgery to date of hospital discharge, up to 3 months
Total hospital charges | From date of index surgery to date of hospital discharge, up to 3 months
Rate of discharge to home | From date of index surgery to date of hospital discharge, up to 3 months
Rate of hospital readmission | 30-day postoperative period
Health-related quality of life | Postoperative (at 30 days)
Receipt of anti-neoplastic therapy | 30-day postoperative period
Overall survival | From date of index surgery to date of death, loss to follow-up, or end of study, whichever comes first, assessed up to 60 months

OTHER OUTCOMES:
Rate of unplanned return to the operating room | 30-day postoperative period
Rate of unplanned hospital readmission | 30-day postoperative period
Rate of hospital readmission | 60-day postoperative period
Rate of hospital readmission | 90-day postoperative period
Health-related quality of life | Postoperative (at 60 days)
Health-related quality of life | Postoperative (at 90 days)
Receipt of anti-neoplastic therapy | 60-day postoperative period
Receipt of anti-neoplastic therapy | 90-day postoperative period
Disease-free survival | From date of index surgery to date of recurrence, death, loss to follow-up, or end of study, whichever comes first, assessed up to 60 months
  In patients who are deemed to have no clinical evidence of disease after the index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nestor F Esnaola, MD, MPH, MBA, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States